CLINICAL TRIAL: NCT05267587
Title: Pre-operative Hypofractionated Stereotactic Radiosurgery for Resectable Brain Metastases
Brief Title: Preop fSRS for Resectable Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21193
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases; Brain Lesion
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Stereotactic Radiosurgery prior to resection (Experimental): Participants will be given hypofractionated stereotactic radiosurgery (fSRS) in 9 Gray Units (Gy) per fraction x 3 consecutive daily fractions (27 Gy total) to the index metastasis that will be resected on Days 1-3 (3 consecutive days). If there are additional non index brain metastasis, they will be treated with standard stereotactic radiosurgery at the time of fSRS. Participants will then undergo stereotactic craniotomy for surgical resection of the index metastasis within 5 days following completion of fSRS.
  Interventions: Radiation: Hypofractionated Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiosurgery — Participants will be given hypofractionated stereotactic radiosurgery (fSRS) in 9 Gray Units (Gy) per fraction x 3 consecutive daily fractions (27 Gy total) to the index metastasis that will be resected.

SUMMARY:
The purpose of the study is to determine whether treatment with pre-operative hypofractionated stereotactic radiosurgery followed by surgery will improve time to local failure (TTLF) compared to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancy other than lymphoma, or germ cell tumor. Brain biopsy is not required unless diagnosis is judged to be in doubt by the treating physician.
* Life expectancy must be deemed to be 3 months or more by a neurosurgeon, radiation oncologist, or medical oncologist with expertise in the treatment of metastatic cancer to the brain.
* Participants must have MRI evidence of >/=1 brain metastasis no less than 10 mm and no greater than 60 mm in maximum diameter, deemed surgically resectable by neurosurgeon, not previously treated with Stereotactic Radiosurgery (SRS) or appropriate for fSRS.
* Each non-index lesion must be </= 4.0 cm in maximal extent on contrasted MRI scan, and not otherwise require resection. The number of non-index lesions allowed will be at the treating physician's discretion, providing the use of whole brain radiotherapy is not used for treatment of these lesions.
* Participants must be either asymptomatic from their brain metastases or have symptoms which are well controlled with steroid medication.
* Systemic therapy such as immunotherapy, targeted therapy, or chemotherapy are permitted at treating physician's discretion.
* Karnofsky Performance Status (KPS) >/=60.
* This study permits the re-enrollment of participant who has discontinued the study due to pre-treatment failure (i.e., the participant has not been treated). If re-enrolled, participant must be re-consented.
* Women of Childbearing Potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to the start of radiation therapy.
* Azoospermic males and WOCBP whoa re continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described.
* Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception (detailed in protocol), which have a failure rate of <1% when used consistently and correctly.

Exclusion Criteria:

* Participants who have germ cell tumors, primary brain tumor, or lymphoma
* Participants with symptoms related to brain metastases not able to be controlled with steroids.
* Women who are pregnant or breastfeeding
* Women of childbearing potential who are not using an effective method of contraception
* Participants deemed medically unfit to undergo surgical resection of brain metastasis by the treating neurosurgeon because of medical comorbidities, such as those who are neurologically or hemodynamically unstable despite appropriate medical interventions.
* Participants who have had whole brain radiation within the previous three months.
* Any prior cranial radiotherapy targeting the index lesion
* Index lesion located in the brainstem
* Any participants with the following imaging findings:

Widespread definitive leptomeningeal metastasis Infratentorial mass effect with fourth ventricle effacement or hydrocephalus Supratentorial mass effect with greater than 10 mm of midline shift or hydrocephalus.

A brain metastasis that is located within 2 mm of the optic chiasm

* Active or prior: documented inherited hypersensitivity syndromes, certain collagen vascular diseases, and certain autoimmune diseases. For example, any radiation hypersensitivity syndrome, including, but not limited to, Gorlin syndrome, multiple sclerosis, ataxia-telangiectasia, scleroderma, and systemic lupus erythematosus.
* Inability to complete MRI with contrast of the brain, or a known allergy to gadolinium
* Participants receiving cytotoxic chemotherapies 7 days prior to or concurrently with fSRS. Note: All other systemic therapies (i.e., molecularly targeted therapies) will be reviewed on a case-by-case basis by study PI to determine if appropriate for study treatment and documented within the research record or EMR.
* If participant's treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved.
* Inability or unwillingness to return for all the required follow-up visits
* Prisoners or individuals who are involuntarily incarcerated
* Individuals who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Time from Start of fSRS until Progression | up to 12 months
  Time from start of hypofractionated stereotactic radiosurgery until first occurrence of local progression of disease, or death. If none of these events occur, patients will be censored on date of last contact.

SECONDARY OUTCOMES:
Time from Start of fSRS until First Development of Leptomeningeal Disease or Death | up to 12 months
  Time from start of hypofractionated stereotactic radiosurgery until first development of leptomeningeal disease, or death. If this event does not occur, patients will be censored on date of last contact.

OTHER OUTCOMES:
Local Control Rate | at 6 months
  Local control rate is defined as the freedom from local progression
Local Control Rate | at 12 months
  Local control rate is defined as the freedom from local progression
Rate of Leptomeningeal Disease (LMD) | at 6 months
  Rate of LMD is defined as the percentage of participants that progressed to leptomeningeal disease
Rate of Leptomeningeal Disease (LMD) | at 12 months
  Rate of LMD is defined as the percentage of participants that progressed to leptomeningeal disease
Rate of distant brain recurrence (DBR) | at 6 months
  Rate of distant brain recurrence defined as the percentage of participants that experienced distant brain recurrence
Rate of distant brain recurrence (DBR) | at 12 months
  Rate of distant brain recurrence defined as the percentage of participants that experienced distant brain recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yu, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States